CLINICAL TRIAL: NCT04922762
Title: Examining the Impact of Exercise Training on Vascular Dysfunction in Individuals With Mental Health Disorders - Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20020955-2
Record Dates: First submitted 2021-05-24; First posted 2021-06-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Vascular Diseases
Keywords: cardiovascular disease; vascular function; PTSD; GAD; Oxidant
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Intensity, Normal Volume Exercise Training (Experimental): Participants will complete study 1 (HM20020955-1) and then 10 weeks of moderate intensity, normal volume exercise training
  Interventions: Behavioral: Moderate Intensity, Normal Volume Exercise Training
- High Intensity, Normal Volume Exercise Training (Experimental): Participants will complete study 1 (HM20020955-1) and then 10 weeks of high intensity, normal volume exercise training
  Interventions: Behavioral: High Intensity, Normal Volume Exercise Training
- Moderate Intensity, High Volume Exercise Training (Experimental): Participants will complete study 1 (HM20020955-1) and then 10 weeks of moderate intensity, high volume exercise training
  Interventions: Behavioral: Moderate Intensity, High Volume Exercise Training

INTERVENTIONS:
Behavioral: Moderate Intensity, Normal Volume Exercise Training — Week 1 3 days/week for 20 minutes/day Performed at 70% of heart rate maximum
  Week 2 3 days/week for 30 minutes/day Performed at 70% of heart rate maximum
  Weeks 3-10 3 days/week for 45 minutes/day Performed at 70% of heart rate maximum
  Arms: Moderate Intensity, Normal Volume Exercise Training
Behavioral: High Intensity, Normal Volume Exercise Training — Week 1 3 days/week for 31 minutes/day 10 minute warm up at 50% of heart rate maximum 2 x 4 minute intervals 4 minutes at 90-95% of heart rate maximum 3 minutes at 70% of heart rate maximum REPEAT 7 minute cool down at 50% of heart rate maximum
  Week 2 3 days/week for 38 minutes/day 10 minute warm up at 50% of heart rate maximum 3 x 4 minute intervals 4 minutes at 90-95% of heart rate maximum 3 minutes at 70% of heart rate maximum REPEAT 2 TIMES 7minute cool down at 50% of heart rate maximum
  Weeks 3-10 3 days/week for 45 minutes/day 10 minute warm up at 50% of heart rate maximum 4 x 4 minute intervals 4 minutes at 90-95% of heart rate maximum 3 minutes at 70% of heart rate maximum REPEAT 3 TIMES 7 minute cool down at 50% of heart rate maximum
  Arms: High Intensity, Normal Volume Exercise Training
Behavioral: Moderate Intensity, High Volume Exercise Training — Week 1 5 days/week for 20 minutes/day Performed at 70% of heart rate maximum
  Week 2 5 days/week for 30 minutes/day Performed at 70% of heart rate maximum
  Weeks 3-10 5 days/week for 45 minutes/day Performed at 70% of heart rate maximum
  Arms: Moderate Intensity, High Volume Exercise Training

SUMMARY:
The purpose of this research study is to examine the effect of various forms of exercise training on blood vessel function in healthy individuals as well as individuals with mental health disorders (posttraumatic stress disorder (PTSD) and/or generalized anxiety disorder (GAD)).

DETAILED DESCRIPTION:
Study #2 is made up of five sessions done on five separate days and the entire study can be completed in as little as 14 weeks. All testing sessions will take place at the Exercise Physiology Research Laboratory. Volunteers will be asked to participate in one initial testing session (Visit 1) lasting < 1 hour that will help make them more familiar with the study equipment and procedures, determine body measures (height, weight, body fat), determine the maximum strength of their forearm and calf, and require one blood draw. The following two testing sessions (Visits 2 and 3) with each session lasting between 2-3 hours that will involve multiple tests designed to determine the health of their blood vessels. For Visit #2 they will be randomly given either antioxidant pills or placebo pills to determine the effect of oxidants on blood vessel health. For Visit #3, they will be given whatever set of pills (antioxidant or placebo) that they did not receive during Visit #2. also include two additional testing days (Visits 5 and 6) that are identical to Visits #2 and #3, two visits to test endurance or strength prior to and after the exercise training (Visit 4 and 7), and ten weeks of exercise training (done 3-5 days per week). The exercise training will include one of three treadmill running programs that differ by exercise intensity and/or exercise frequency.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy and free of overt cardiovascular, pulmonary, or metabolic disease
* for PTSD group, a score of ≥ 33 on PCL-5 checklist
* for GAD group, a score of ≥ 10 on the GAD-7 self-report scale and < 33 on the PCL-5 checklist
* for Healthy Control group, a score of ≤ 10 on the GAD-7 self-report scale and < 33 on the PCL-5 checklist

Exclusion Criteria:

* taking medications that could influence cardiovascular function
* current smokers who have recently quit smoking
* illicit drug use or excessive alcohol consumption
* pregnant women
* significant calorie restriction or vitamin/mineral deficiencies
* limited English proficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arm Vascular Function at Rest (Flow Mediated Dilation Test) | Baseline to the end of the final visit, about 14 weeks
  Change in Brachial Artery Dilation from Baseline Values
Leg Vascular Function (Passive Leg Movement Test) | Baseline to the end of the final visit, about 14 weeks
  Change in Leg Blood Flow Values from Baseline
Arm Vascular Function in Response to Exercise (Handgrip Exercise Test) | Baseline to the end of the final visit, about 14 weeks
  Change in Brachial Artery Dilation from Baseline Values

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Garten, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States